CLINICAL TRIAL: NCT06775834
Title: Safety and Pharmacokinetic Study of HRS-1893 Tablets in Subjects With Mild and Moderate Renal Insufficiency and Healthy Subjects
Brief Title: Safety and Pharmacokinetics Study of HRS-1893 Tablets in Healthy Subjects and Those With Impaired Kidney Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shandong Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HRS-1893-103
Record Dates: First submitted 2025-01-09; First posted 2025-01-15 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Hypertrophic Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Normal Renal Function Group (Experimental)
  Interventions: Drug: HRS-1893
- Mild Renal Impairment Group (Experimental)
  Interventions: Drug: HRS-1893
- Moderate Renal Impairment Group (Experimental)
  Interventions: Drug: HRS-1893

INTERVENTIONS:
Drug: HRS-1893 — HRS-1893 tablets.

SUMMARY:
The primary objective is to evaluate pharmacokinetics of HRS-1893 tablets in subjects with impaired kidney function in comparison with healthy subjects, to develop dose recommendations for patients with renal impairment.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent before the trial, and fully understand the content, process and possible adverse reactions of the trial;
2. Male or female subjects aged 18 to 65 (including 18 and 65);
3. Body mass index (BMI) ranges from 19 kg/m2 to 28 kg/m2 (including 18 and 28);
4. The glomerular filtration rate should meet the following criteria (GFR, mL/min): Subjects with mild renal impairment: 60-89 mL/min; Subjects with moderate renal impairment: 30-59 mL/min.

Exclusion Criteria:

1. Suspected allergy to the study drug or any component of the study drug;
2. Patients with cardiogenic shock, severe conduction block, sick sinus syndrome, heart failure, sustained tachyarrhythmia, torsades de pointes (Tdp) or ventricular tachycardia, history of clinically significant T wave changes, myocardial infarction, angina pectoris;
3. People with conditions associated with reduced neuromuscular transmission (myasthenia gravis, Lambert-Eaton syndrome, Duchenne muscular dystrophy);
4. Patients with a history of gastric or intestinal surgery that may affect drug absorption;
5. Participants with renal insufficiency who were judged by the investigator to be ineligible for the study;
6. Patients with large fluctuations or rapid deterioration of renal function within 2 weeks before administration, as judged by the investigator;
7. Subjects receiving renal replacement therapy within 3 months of the screening period or during the expected trial period;
8. Within 3 months before screening, patients with underlying diseases that induced chronic kidney disease and were poorly controlled according to the investigator's evaluation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2025-02-11 (Actual); Primary Completion 2025-07-23 (Actual); Study Completion 2025-07-23 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) | 0 hour to 16 days after the dosing.
Area under the plasma concentration-time curve from time zero to the time of last quantifiable analyte concentration (AUC0-t) | 0 hour to 16 days after the dosing.
Area under the plasma concentration-time curve from time zero extrapolated to infinity (AUC0-∞) | 0 hour to 16 days after the dosing.

SECONDARY OUTCOMES:
Time to reach maximum plasma concentration (Tmax) | 0 hour to 16 days after the dosing.
Terminal half-life (t1/2) | 0 hour to 16 days after the dosing.
Apparent clearance (CL/F) | 0 hour to 16 days after the dosing.
Apparent volume of distribution (Vz/F) | 0 hour to 16 days after the dosing.
Cumulative excretion (Ae) | 0 hour to 16 days after the dosing.
Plasma protein binding rate (PPB) | 0 hour to 16 days after the dosing.
Incidence and severity of adverse events (AEs) | 0 hour to 16 days after the dosing.

CONTACTS AND LOCATIONS:
Locations (1):
- Sichuan Provincial People's Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided